Participant ID: EA\_\_\_\_

London



## **CONSENT FORM**

Study Protocol number: 14SM2070

Full Title of Project: THE IMPACT OF AGE ON ADAPTIVE IMMUNITY IN ADULTS INFECTED

WITH RESPIRATORY SYNCYTIAL VIRUS Principal investigator: Professor Christopher Chiu

| | | Please | initial |
|---|---|---|---|
| 1. | I confirm that I have read and understand the participant information sheet <b>Version XX dated XXXXXXXXX</b> for the above study and have had the opportunity to ask questions which have been answered fully. | | |
| 2. | I understand that my participation is voluntary, and I am free to withdraw at any time, without giving any reason and without my legal rights nor treatment / healthcare being affected. | | |
| 3. | I understand that sections of any of my medical notes may be looked at by responsible individuals from Imperial College, Imperial College Healthcare NHS Trust or from regulatory authorities, where it is relevant to my taking part in this research. | | |
| 4. | I understand that, after having my medical history taken, a physical examination, Chest X-ray, urine, breathing and blood tests will make sure I am eligible, I will be enrolled to be inoculated with RSV. | | |
| 5. | I understand that I will undergo four bronchoscopies as part of this study. | | |
| 6 | After inoculation with RSV, I agree to remain in the residential facility at all times for a period of 8-10 nights during the study. | | |
| 7. | I am willing to be housed in a mixed-gender ward during the residential period. | Yes | No |
| 8. | <b>OPTIONAL</b> - I give consent for information collected about me to be used to support other research or in the development of a new test, medication, medical device or treatment (delete as applicable) by an academic institution or commercial company in the future, including those outside of the United Kingdom (which Imperial has ensured will keep this information secure). | Yes | No |
| 9. | <b>OPTIONAL</b> - I give consent for samples (human tissue) collected about me to be used to support other research or in the development of a new test, medication, medical device or treatment (delete as applicable) by an academic institution or commercial company in the future, including those outside of the United Kingdom (which Imperial has ensured will keep this information secure). | Yes | No |
| 10. | I understand that tissue samples and / or data collected from me are a gift donated to Imperial College and that I will not personally benefit financially if this research leads to an invention and/or the successful development of a new test, medication treatment, product or service. | | |
| 11. | I agree to my General Practitioner being informed of my participation in the study, and the request of my past medical history. | | |
| 12. | The results of some study measurements of my immune response might warrant further investigation to assess the correlation between the immune response and some genetic characteristics. OPTIONAL - I agree to my tissue samples being used to undertake genetic research which may have the potential to generate data that can be tracked back to me | Yes | No |

| Participant ID: EA | Imperial College | Imperial College Healthcare | NHS |
|--------------------|------------------|-----------------------------|-----|
| | London | NHS Trust | |

| 13. | <b>OPTIONAL</b> - I give / do not give (delete/mark as applicable) consent to being contacted about the possibility to take part in other research studies. | Yes | No |
|---|---|---|---|
| 14. | I consent to take part in "THE IMPACT OF AGE ON ADAPTIVE IMMUNITY IN ADULTS INFECTED WITH RESPIRATORY SYNCYTIAL VIRUS" (INFLAMMAGE) Study | | · |

| Participant |
|--------------|
| Full Name |
| Signature |
| Date |
| Investigator |
| Full Name |
| Signature |
| Date |

1 copy for participant; 1 copy for Principal Investigator; 1 copy to be kept with hospital notes